CLINICAL TRIAL: NCT00001245
Title: Study of Patients With Known or Suspected Infection With Strongyloides Stercoralis
Brief Title: Study of Patients With Strongyloides Stercoralis Infection
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 890174; 89-I-0174
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-05

CONDITIONS: HIV Infection; Nematode Infection; Strongyloidiasis
Keywords: Strongyloidiasis; Immediate Hypersensitivity Skin Test; IgE; Nematode; Immunosuppression; Skin Test; Diagnosis; Intestinal Helminth; Immediate Hypersensitivity
MeSH Terms: conditions — HIV Infections; Nematode Infections; Strongyloidiasis; Enterobiasis; Disease; Hypersensitivity, Immediate

SUMMARY:
This study will explore faster and easier ways to detect infection with the intestinal parasite Strongyloides stercoralis and learn more about the conditions under which it causes serious disease. Ordinarily, the Strongyloides helminth (type of intestinal worm) causes only few, if any, symptoms, but in people with weakened immunity it may be very serious, and even deadly.

People between 5 and 80 years of age with known or suspected S. stercoralis infection, or infection with another helminth, such as filariasis, that might cause a cross-reaction with S. stercoralis may be eligible for this study.

Participants found to be infected with S. stercoralis will be treated with ivermectin, thiabendazole, or albendazole. In addition, they will undergo the following tests and procedures:

* Blood tests and stool samples: Samples will be collected before and after treatment to check general health status and immune function, and to look for parasites in stool. Up to 50 milliliters (10 teaspoons) of blood will be drawn in adults and up to 25 ml (5 teaspoons) in children.
* Skin tests: A test similar to those used for tuberculosis and allergies will be conducted to determine if there is sensitization to products of the parasite. Such a test might be used as a rapid method to diagnose the infection. About three drops of several different antigens (proteins) are injected into the skin of the arm. After 15 to 20 minutes, the area is checked to see if a red spot has formed and, if so, the spot is measured.

DETAILED DESCRIPTION:
This study is directed to patients with known or suspected Strongyloides stercoralis infection because it is a relatively common parasitic infection, even in the United States. It is difficult to diagnose, and efficacy of treatment is difficult to evaluate. Some infected individuals can develop serious even fatal, disease under certain conditions of immunosuppression. Because newer diagnostic methods are needed to diagnose this infection, we have developed new diagnostics that will be evaluated in comparison to more standard diagnostic tests. Serum and cells will also be collected from patients on this protocol to understand the cellular and humoral response to the parasite and its antigens. All subjects proven to have Strongyloides stercoralis infection will be treated with standard therapy and followed to assess both the efficacy of treatment and the changes in humoral and cellular immune responses induced by treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age of 5 to 80 years and of either sex.

Access to primary medical care provider outside of the NIH

Ability to give written informed consent (for adults) and parental consent (for those under 18)

Presence of known or suspected infection with Stronglyloides stercoralis, such as significant peripheral blood eosinophilia (greater than 1000 eosinophils/mm(3)) for which no other cause is apparent.

Willingness to participate and provide blood for in vitro assays and serum storage.

EXCLUSION CRITERIA:

Less than 5 years of age

Pregnancy is not a criterion for exclusion.

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 650
Dates: Start 1989-08; Primary Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Neva FA. Biology and immunology of human strongyloidiasis. J Infect Dis. 1986 Mar;153(3):397-406. doi: 10.1093/infdis/153.3.397. PMID 3081656
- [Background] Newton RC, Limpuangthip P, Greenberg S, Gam A, Neva FA. Strongyloides stercoralis hyperinfection in a carrier of HTLV-I virus with evidence of selective immunosuppression. Am J Med. 1992 Feb;92(2):202-8. doi: 10.1016/0002-9343(92)90113-p. PMID 1543206
- [Background] Sato Y, Otsuru M, Takara M, Shiroma Y. Intradermal reactions in strongyloidiasis. Int J Parasitol. 1986 Feb;16(1):87-91. doi: 10.1016/0020-7519(86)90070-6. No abstract available. PMID 3699981
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_1989-I-0174.html